CLINICAL TRIAL: NCT03687619
Title: The Effects of Cognitive Orientation to Daily Occupational Performance and Conductive Education Approaches on Fine Motor Skills, Activity and Participation Limitations in Children With Down Syndrome: Randomized Controlled Trial
Brief Title: Cognitive Orientation to Daily Occupational Performance and Conductive Education Approaches on Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Hülya Özbeşer, PT. Ms, Eastern Mediterranean University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ETK00-218-0213
Record Dates: First submitted 2018-09-26; First posted 2018-09-27 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Down Syndrome, Trisomy 21
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CO-OP (Experimental): Cognitive Orientation to daily Occupational Performance (CO-OP) is a top-down approach. This programme will be conducted as a small group. Each group will averagely have 5 children. The primary investigator will conduct the programmes. It will be one hour session, twice a week, 12 weeks.
  Interventions: Other: CO-OP
- Conductive Education (Experimental): Conductive Education is a down-top approach. This programme will be conducted as a small group. Each group will averagely have 5 children. The primary investigator will conduct the programmes. It will be one hour session, twice a week, 12 weeks.
  Interventions: Other: Conductive Education

INTERVENTIONS:
Other: CO-OP — Interventions (from top to down) related to the development of fine-motor skills
  Arms: CO-OP
Other: Conductive Education — Interventions (from down to top) related to the development of fine-motor skills
  Arms: Conductive Education

SUMMARY:
This study will be conducted to investigate and compare the effects of Cognitive Orientation to Daily Occupational Performance (CO-OP) and Conductive Education (CE) on fine motor skills, activity, and participation limitations in children with DS. Children with DS aged 7-18 years will be included. Both CO-OP and CE interventions will last 12 weeks and be conducted for 2 sessions per week in the cross-over randomized study. Following 12-week wash-out period, interventions will be changed for each group.

DETAILED DESCRIPTION:
Down syndrome (DS) is a chromosomal anomaly characterized by the presence of an extra copy of genetic material on the 21st chromosome. Sensory, motor, cognitive and perceptual impairments can be seen in children with DS. These impairments probably affect the development and learning of their various fundamental and complex actions. Those children experience decreased motor proficiency, reduced social participation and lower life quality.

Fine motor skills are important for children's everyday functioning such as dressing, feeding, bathing, holding objects, cutting etc. In addition, fine motor skills are related to cognitive, social and academic abilities in children.

This study will be conducted to investigate and compare the effects of Cognitive Orientation to Daily Occupational Performance (CO-OP) and Conductive Education (CE) on fine motor skills, activity, and participation limitations in children with DS. Children with DS aged 7-18 years will be included.

Random allocation software will be used to assign CO-OP or CE to participants. Both CO-OP and CE interventions will last 12 weeks and be conducted for 2 sessions per week. Both intervention will be applied as groups including 3-4 children. Following 12-week wash-out period, interventions will be changed for each group. Two meetings before and during the study will be done in order to inform parents about the interventions and their effects. Another investigator who is blind about the groups will conduct the assessments before and after both first and second treatment durations so 4 assessments will be done in total. At the end of whole treatment schedule, a satisfaction form will be asked from the parents for feedback about both interventions.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 7 and 18 years
* Children who can understand cognitive skills given and can verbally communicate
* Children who can specify at least 3 activities
* Children who have adequate motivation

Exclusion Criteria:

* Caregivers or parents who have inadequate cognitive levels for the study progression
* Children who participate in any physiotherapy/ergo-therapy schedules for at least 3 months
* Children who have Cognitive Orientation to daily Occupational Performance and Conductive Education program.
* Children who have other neurological problems (except Down Syndrome)
* Children who have undergone orthopedic surgery related to upper limbs
* Children who have other health and behavioral problems which can affect the participation in the study

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2019-12-22 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
performance quality rating scale | 12 weeks
  The PQRS rates performance quality on a 10-point scale, with a score of 1 indicating ''can't do the skill at all'' and 10 indicating ''does the skill very well''. An independent observer rates performances from video recorded trials of each skill at all assessment points.

SECONDARY OUTCOMES:
Nine Hole Peg Test | 12 weeks
  The Nine-Hole Peg Test is a timed dexterity test that evaluates the ability to pick up nine 1¼-inch-long plastic pegs from a shallow dish, place them one at a time into a pegboard, and remove them one at a time back into the dish. The total time to complete the task for each hand will be recorded in seconds.
Bruininks-Oseretsky Motor Proficiency Test - Brief Form | 12 weeks
  It will be used to determine the motor skills of the children. Bilateral coordination, balance, strength and speed-agility will be measured to specify gross motor skills, while fine motor precision, fine motor integration, manual dexterity, and upper limb coordination will be measured for fine motor skills.
Canadian Occupational Performance Measure | 12 weeks
  The COPM is an outcome measure that, through a semi-structured interview, is designed to (a) identify and prioritize occupational performance issues or goals, and (b) measure clients' self perceived changes in occupational performance and satisfaction with their performance over time, of identified goals.
Dynamic Performance Analysis | 12 weeks
  DPA is a dynamic, iterative process, carried out as the client performs the occupation. The purpose of DPA is to identify where performance breaks down and test out solutions.This analysis will be used within the concept of CO-OP.
Child Health Questionnaire- Parent Form | 12 weeks
  The CHQ PF-50 is a 50 item, parent-completed questionnaire designed to measure the physical and psychosocial well-being of children with and without chronic conditions. Reliability and validity of Turkish version have been shown. The CHQ PF-50 measures components of physical and psychosocial functioning in 12 categories (subscales). The subscales used for our analyses included: physical functioning, role/social limitations (note: we call this subscale "School & Friends" since it measures the degree to which schoolwork or activities with friends are limited due to problems with physical health), bodily pain/ discomfort, mental health, and self-esteem.
Goal Attainment Scaling | 12 weeks
  The goal attainment scale is characterised by five levels of achievement. The expected outcome is the middle or 'zero' score. This expected outcome is determined first and then two better and two worse outcomes are documented. It enables individualised goals to be set and allows measurement of clinically important change which may not be detected by standardised assessments
Parent Satisfaction Form | 12 weeks
  It is a semi-structured questionnaire which will indicate the satisfaction level of parents from both approaches.

CONTACTS AND LOCATIONS:
Overall Officials: Emine H. Tüzün, Prof. Dr., Principal Investigator — Instructor; Hülya Özbeşer, MSc. PT, Principal Investigator — Instructor; Levent Eker, M. D., Principal Investigator — Instructor
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus